CLINICAL TRIAL: NCT00098150
Title: A Follow-Up Study of Patients Previously Treated in a Core Study With Pimecrolimus Tablets for Atopic Dermatitis
Brief Title: Follow-Up Study of Patients Previously Treated With Pimecrolimus Tablets for Atopic Dermatitis
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Other Study IDs: Ext 1 to ASM981C202
Record Dates: First submitted 2004-12-03; First posted 2004-12-06 (Estimated); Last update posted 2006-08-31 (Estimated); Status verified 2006-08

CONDITIONS: Atopic Dermatitis
Keywords: Safety, atopic dermatitis, adverse event, SAE, extension
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
This extension study is being conducted to collect post-treatment safety information on patients who previously participated in the core clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients who participated in the core clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66
Dates: Start 2004-07